CLINICAL TRIAL: NCT00460044
Title: Plasma ADMA Concentrations at Birth and Mechanical Ventilation in Preterm Infants
Brief Title: ADMA and Mechanical Ventilation in Preterm Infants
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Other Study IDs: HK0607
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Last update posted 2007-04-13 (Estimated); Status verified 2007-04

CONDITIONS: Premature Birth
Keywords: ADMA; Preterms; infants; mechanical ventilation; Preterm infants
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to study the relation between mechanical ventilation and ADMA concentrations at birth.

DETAILED DESCRIPTION:
Nitric oxide (NO) plays an important role in the normal development and maturation of the lungs. In addition, NO is an important mediator of vascular smooth muscle relaxation, ventilation perfusion matching, neurotransmission and host defence and bacteriostasis. Asymmetric dimethylarginine (ADMA) is an endogenous derivative of arginine that inhibits NOS and thereby the bioavailability of NO. Preterm infants have increased concentrations of ADMA. Therefore, inhibition of NO by increased concentrations of ADMA which could be associated with reduced pulmonary functioning.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age < 32 weeks
* Birth weight < 1500 gram
* Written informed consent of parents

Exclusion Criteria:

* Congenital abnormalities
* Chromosomal abnormalities

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35
Dates: Start 2002-01; Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R M van Elburg, MD, PhD, Study Director — Amsterdam UMC, location VUmc